CLINICAL TRIAL: NCT02337946
Title: A Phase 2 Randomized Study Comparing the Efficacy and Safety of mFOLFOX6+Panitumumab Combination Therapy and 5-FU/LV+Panitumumab Combination Therapy in the Patients With Chemotherapy-Naive Unresectable Advanced Recurrent Colorectal Carcinoma of KRAS Wild-Type After 6 Cycles of Combination Therapy With mFOLFOX6+Panitumumab
Brief Title: Safety and Efficacy Study of mFOLFOX6 + Panitumumab Combination Therapy and 5-FU/LV + Panitumumab Combination Therapy in Participants With Chemotherapy-naïve Unresectable Advanced Recurrent Colorectal Carcinoma
Acronym: SAPPHIRE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Panitumumab-2003; U1111-1161-8871 (Registry Identifier: UTN (WHO)); 183/NRP-005 (Other: Secondary Takeda ID); JapicCTI-142668 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2014-09-30; First posted 2015-01-14 (Estimated); Results first posted 2019-03-01 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-08

CONDITIONS: Colorectal Carcinoma
Keywords: Metastatic colorectal cancer, Panitumumab, mFOLFOX6, First-line
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Oxaliplatin; Fluorouracil; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Panitumumab (Pmab) 6 mg/kg, intravenous drip infusion (DIV), at Day 1, oxaliplatin (OXA) 85 mg/m^2, DIV, at Day 1, levofolinate (l LV) 200 mg/m^2, DIV, at Day 1, fluorouracil (5-FU) 400 mg/m^2, intravenous (IV) at Day 1, 5-FU 2400 mg/m^2, continuous intravenous infusion (CIV), at Day 2 once every two weeks from cycle 1 through cycle 6 as protocol treatment 1 followed by Pmab 6 mg/kg, DIV, at Day 1, OXA 85 mg/m^2, DIV, at Day 1, l LV 200 mg/m^2, DIV, at Day 1, 5-FU 400 mg/m^2, IV, at Day 1, 5-FU 2400 mg/m^2, CIV, at Day 2 once every two weeks from cycle 7 until progressive disease or intolerance.
  Interventions: Drug: oxaliplatin (OXA), levofolinate calcium (l-LV), 5-FU, panitumumab
- Group B (Experimental): Pmab 6 mg/kg, DIV, at Day 1, OXA 85 mg/m^2, DIV, at Day 1, l LV 200 mg/m^2, DIV, at Day 1, 5-FU 400 mg/m^2, IV, at Day 1, 5-FU 2400 mg/m^2, CIV, at Day 2 once every two weeks from cycle 1 through cycle 6 as protocol treatment 1 followed by Pmab 6 mg/kg, DIV, at Day 1, l LV 200 mg/m^2, DIV, at Day 1, 5-FU 400 mg/m^2, IV, at Day 1, 5-FU 2400 mg/m^2, CIV, at Day 2 once every two weeks from cycle 7 until progressive disease or intolerance.
  Interventions: Drug: oxaliplatin (OXA), levofolinate calcium (l-LV), 5-FU, panitumumab

INTERVENTIONS:
Drug: oxaliplatin (OXA), levofolinate calcium (l-LV), 5-FU, panitumumab — oxaliplatin (OXA), levofolinate calcium (l-LV), panitumumab: intra-venous infusion 5-FU: bolus and continuous intra-venous infusion
  Arms: Group A
Drug: oxaliplatin (OXA), levofolinate calcium (l-LV), 5-FU, panitumumab
  Arms: Group B

SUMMARY:
The purpose of this study is to exploratorily examine efficacy and safety in the participants with chemotherapy-naïve unresectable, advanced/recurrent colorectal carcinoma of Kirsten rat sarcoma-2 virus (KRAS) wild-type who have been treated with 6 cycles (2 weeks/cycle) of first-line mFOLFOX6 + panitumumab combination therapy and then assigned to two groups i.e., a group receiving 5-FU/LV + panitumumab combination therapy and a group receiving mFOLFOX6 + panitumumab combination therapy.

DETAILED DESCRIPTION:
The drug being tested in this study is called panitumumab. Panitumumab is being tested to treat people who have advanced/recurrent colorectal carcinoma of KRAS wild-type. This study will look at the efficacy and safety of 5-FU/LV + panitumumab(Pmab) combination therapy or mFOLFOX6 + Pmab combination therapy in the participants.

The study will enroll 164 patients. All participants will receive 6 cycles of Protocol Treatment [1]: Pmab 6 mg/kg, DIV, at Day 1, OXA 85 mg/m^2, DIV, at Day 1, l LV 200 mg/m^2, DIV, at Day 1, 5-FU 400 mg/m^2, IV, at Day 1, 5-FU 2400 mg/m^2, CIV, at Day 2 once every two weeks from cycle 1 through cycle 6.

Then they will be randomly assigned (by chance, like flipping a coin) to one of the treatment groups.

* Group A
* Group B

This multi-center trial will be conducted in Japan. The overall time to participate in this study is approximately 20 months.

ELIGIBILITY:
Inclusion Criteria for enrollment:

1. Participants with unresectable adenocarcinoma originating in the large intestine (excluding carcinoma of the appendix and anal canal cancer)
2. Participants with measurable lesion(s) according to the RECIST ver. 1.1
3. Participants who have not received chemotherapy for colorectal cancer. Participants who experience relapse more than 6 months after the final dose of perioperative adjuvant chemotherapy with fluoropyrimidine agents may be enrolled.
4. Aged ≥ 20 years at the time of enrollment
5. Participants classified as KRAS wild-type. However, the criteria will be changed to all patients who are verified to be of KRAS and NRAS wild-type when the KRAS and NRAS tests come to be covered by National Health Insurance, and the tests become feasible at medical institutions.
6. Participants who satisfy the following criteria for the major organ function in tests performed within 14 days prior to enrollment

   1. Neutrophil count ≥ 1.5 × 10^3/μL
   2. White blood cell count ≥ 3.0 × 10^3/μL
   3. Platelet count ≥ 10.0 × 10^4/μL
   4. Hemoglobin ≥ 9.0 g/dL
   5. Total bilirubin ≤ 2.0 mg/dL
   6. AST ≤ 100 U/L (≤ 200 U/L if liver metastases are present)
   7. ALT ≤ 100 U/L (≤ 200 U/L if liver metastases are present)
   8. Serum creatinine ≤ 1.5 mg/dL
7. Participants who are assessed at Eastern Cooperative Oncology Group (ECOG) performance status (P.S.) of 0 or 1
8. Life expectancy of ≥ 6 months after enrollment
9. Participants who have given written consent to take part in the study after detailed explanation of the study prior to enrollment

Inclusion criteria for randomization:

1. Participants who have received 6 cycles of mFOLFOX6 + panitumumab combination therapy
2. Participants who are assessed at ECOG P.S. of 0-1 in the 6th cycle.
3. Participants for whom PD or not evaluable has been denied on the RECIST 1.1 based on imaging tests conducted after the day of administration in the 6th cycle within 14 days (2 weeks).

Exclusion Criteria for enrollment:

1. Radiotherapy received for a measurable lesion
2. Radiotherapy received within 28 days (4 weeks) prior to enrollment for a lesion other than measurable lesions. However, treatment to relieve pain associated with metastatic bone tumors was allowed.
3. Known brain metastasis or strongly suspected of brain metastasis
4. Synchronous cancers or metachronous cancers with a disease-free period of ≤ 5 years (excluding colorectal cancer) excluding mucosal cancers cured or be possibly cured by regional resection (esophageal, stomach, and cervical cancer, non-melanoma skin cancer, bladder cancer, etc.).
5. Body cavity fluid that requires treatment (pleural effusion, ascites, pericardial effusion, etc.)
6. Participants who do not want to use contraception to prevent pregnancy, and women who are pregnant or breast-feeding, or test positive for pregnancy
7. Active hemorrhage requiring blood transfusion
8. Disease requiring systemic steroids for treatment (excluding topical steroids)
9. Intestinal resection and colostomy within 2 weeks prior to enrollment
10. History or obvious and extensive CT findings of interstitial pulmonary disease (interstitial pneumonia, pulmonary fibrosis, etc.)
11. Serious drug hypersensitivity
12. Local or systemic active infection requiring treatment, or fever indicating infection
13. Intestinal paralysis, gastrointestinal obstruction, or uncontrollable diarrhea (incapacitating symptoms despite adequate treatment)
14. Active hepatitis B and/or active hepatitis C
15. Known human immunodeficiency virus infection
16. Other patients judged by the investigator or subinvestigator to be ineligible for enrollment in the study

Exclusion criteria for randomization:

1. Participants in whom interstitial pneumonia has been newly diagnosed during the period from registration to randomization
2. Participants who have received radiotherapy during the period from registration to randomization
3. Other Participants judged by the investigator or sub-investigator to be ineligible for enrollment in the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2014-10-16 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (49):
- Japan (49):
  - Nagakute, Aichi-ken
  - Nagoya, Aichi-ken
  - Okazaki, Aichi-ken
  - Toyoaki, Aichi-ken
  - Yachiyo, Chiba
  - Kitakyushu, Fukuoka
  - Tagawa, Fukuoka
  - Aizu-Wakamatsu, Fukushima
  - Kakamigahara, Gifu
  - Tajimi, Gifu
  - Hakodate, Hokkaido
  - Kushiro, Hokkaido
  - Amagasaki, Hyōgo
  - Kakogawa, Hyōgo
  - Kobe, Hyōgo
  - Nishinomiya, Hyōgo
  - Kahoku, Ishikawa-ken
  - Kanazawa, Ishikawa-ken
  - Morioka, Iwate
  - Kida-gun, Kagawa-ken
  - Marugame, Kagawa-ken
  - Takamatsu, Kagawa-ken
  - Kawasaki, Kanagawa
  - Yokohama, Kanagawa
  - Nangoku, Kochi
  - Sendai, Miyagi
  - Matsumoto, Nagano
  - Suwa, Nagano
  - Sasebo, Nagasaki
  - Higashiosaka, Osaka
  - Hirakata, Osaka
  - Izumi, Osaka
  - Izumisano, Osaka
  - Sakai, Osaka
  - Tondabayashi, Osaka
  - Hidaka, Saitama
  - Izumo, Shimane
  - Fujioka, Shizuoka
  - Shimonoseki, Yamaguchi
  - Akita
  - Fukui
  - Fukuoka
  - Gifu
  - Hiroshima
  - Kyoto
  - Nagasaki
  - Okinawa
  - Osaka
  - Saga

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- [Background] Munemoto Y, Nakamura M, Takahashi M, Kotaka M, Kuroda H, Kato T, Minagawa N, Noura S, Fukunaga M, Kuramochi H, Touyama T, Takahashi T, Miwa K, Satake H, Kurosawa S, Miura T, Mishima H, Sakamoto J, Oba K, Nagata N. SAPPHIRE: a randomised phase II study of planned discontinuation or continuous treatment of oxaliplatin after six cycles of modified FOLFOX6 plus panitumumab in patients with colorectal cancer. Eur J Cancer. 2019 Sep;119:158-167. doi: 10.1016/j.ejca.2019.07.006. Epub 2019 Aug 21. PMID 31445198
- [Derived] Nagata N, Mishima H, Kurosawa S, Oba K, Sakamoto J. mFOLFOX6 Plus Panitumumab Versus 5-FU/LV Plus Panitumumab After Six Cycles of Frontline mFOLFOX6 Plus Panitumumab: A Randomized Phase II Study of Patients With Unresectable or Advanced/Recurrent, RAS Wild-type Colorectal Carcinoma (SAPPHIRE)-Study Design and Rationale. Clin Colorectal Cancer. 2017 Jun;16(2):154-157.e1. doi: 10.1016/j.clcc.2017.02.001. Epub 2017 Mar 1. PMID 28284575

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 72 investigative sites in Japan from 16 October 2014 to 31 March 2017 (as Primary Completion Date). After that, overall study completion of this study was occurred on 31 August 2017.
Pre-assignment Details: Participants with a diagnosis of colorectal carcinoma were enrolled to receive protocol treatment (1) up to cycle 6 followed by randomization, received 1 out of 2 treatments from protocol treatment (2) group A and group B.
Groups:
- Protocol Treatment 1: Panitumumab (Pmab) 6 mg/kg, intravenous drip infusion (DIV), at Day 1, oxaliplatin (OXA) 85 mg/m^2, DIV, at Day 1, levofolinate (l LV) 200 mg/m^2, DIV, at Day 1, fluorouracil (5-FU) 400 mg/m^2, intravenous (IV) at Day 1, 5-FU 2400 mg/m^2, continuous intravenous infusion (CIV), at Day 2 once every two weeks from cycle 1 through cycle 6 as protocol treatment 1.
- Protocol Treatment Period 2: Group A: Panitumumab (Pmab) 6 mg/kg, intravenous drip infusion (DIV), at Day 1, oxaliplatin (OXA) 85 mg/m^2, DIV, at Day 1, levofolinate (l LV) 200 mg/m^2, DIV, at Day 1, fluorouracil (5-FU) 400 mg/m^2, intravenous (IV) at Day 1, 5-FU 2400 mg/m^2, continuous intravenous infusion (CIV), at Day 2 once every two weeks from cycle 1 through cycle 6 as protocol treatment 1 followed by Pmab 6 mg/kg, DIV, at Day 1, OXA 85 mg/m^2, DIV, at Day 1, l LV 200 mg/m^2, DIV, at Day 1, 5-FU 400 mg/m^2, IV, at Day 1, 5-FU 2400 mg/m^2, CIV, at Day 2 once every two weeks from cycle 7 until progressive disease or intolerance.
- Protocol Treatment Period 2: Group B: Pmab 6 mg/kg, DIV, at Day 1, OXA 85 mg/m^2, DIV, at Day 1, l LV 200 mg/m^2, DIV, at Day 1, 5-FU 400 mg/m^2, IV, at Day 1, 5-FU 2400 mg/m^2, CIV, at Day 2 once every two weeks from cycle 1 through cycle 6 as protocol treatment 1 followed by Pmab 6 mg/kg, DIV, at Day 1, l LV 200 mg/m^2, DIV, at Day 1, 5-FU 400 mg/m^2, IV, at Day 1, 5-FU 2400 mg/m^2, CIV, at Day 2 once every two weeks from cycle 7 until progressive disease or intolerance.
Period: Protocol Treatment 1 Period
Arm/Group | Protocol Treatment 1 | Protocol Treatment Period 2: Group A | Protocol Treatment Period 2: Group B
Started | 164 | 0 | 0
Completed | 114 | 0 | 0
Not Completed | 50 | 0 | 0
Not completed — Adverse Event | 7 | 0 | 0
Not completed — Major Protocol Deviation | 1 | 0 | 0
Not completed — Voluntary Withdrawal | 6 | 0 | 0
Not completed — Lack of Efficacy | 15 | 0 | 0
Not completed — Death During Protocol Treatment | 3 | 0 | 0
Not completed — Surgery Aimed at Curative Resection | 9 | 0 | 0
Not completed — Did not Meet Entrance Criteria | 1 | 0 | 0
Not completed — Reason not specified | 8 | 0 | 0
Period: In-between Period
Arm/Group | Protocol Treatment 1 | Protocol Treatment Period 2: Group A | Protocol Treatment Period 2: Group B
Started | 114 | 0 | 0
Completed | 113 | 0 | 0
Not Completed | 1 | 0 | 0
Not completed — Without Informed Consent | 1 | 0 | 0
Period: Protocol Treatment 2 Period
Arm/Group | Protocol Treatment 1 | Protocol Treatment Period 2: Group A | Protocol Treatment Period 2: Group B
Started | 0 | 56 | 57
Safety Population | 0 | 56 | 54
Completed | 0 | 5 | 7
Not Completed | 0 | 51 | 50
Not completed — Adverse Event | 0 | 9 | 9
Not completed — Voluntary Withdrawal | 0 | 3 | 1
Not completed — Lack of Efficacy | 0 | 29 | 29
Not completed — Death During Protocol Treatment | 0 | 1 | 0
Not completed — Surgery Aimed at Curative Resection | 0 | 5 | 7
Not completed — Reason not specified | 0 | 4 | 4

BASELINE CHARACTERISTICS:
Population: Enrolled participants included all participants who were enrolled and received protocol treatment 1.
Groups:
- Entire Study Population: Participants who received Panitumumab (Pmab) 6 mg/kg, intravenous drip infusion (DIV), at Day 1, oxaliplatin (OXA) 85 mg/m^2, DIV, at Day 1, levofolinate (l LV) 200 mg/m^2, DIV, at Day 1, fluorouracil (5-FU) 400 mg/m^2, intravenous (IV) at Day 1, 5-FU 2400 mg/m^2, continuous intravenous infusion (CIV), at Day 2 once every two weeks from cycle 1 through cycle 6 as protocol treatment 1 followed by either Pmab 6 mg/kg, DIV, at Day 1, OXA 85 mg/m^2, DIV, at Day 1, l LV 200 mg/m^2, DIV, at Day 1, 5-FU 400 mg/m^2, IV, at Day 1, 5-FU 2400 mg/m^2, CIV, at Day 2 once every two weeks from cycle 7 until progressive disease or intolerance or Pmab 6 mg/kg, DIV, at Day 1, l LV 200 mg/m^2, DIV, at Day 1, 5-FU 400 mg/m^2, IV, at Day 1, 5-FU 2400 mg/m^2, CIV, at Day 2 once every two weeks from cycle 7 until progressive disease or intolerance.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 164
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 109
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Japan | 164
Histological Type of Adenocarcinoma [Count of Participants; unit: Participants]
  Well differentiated adenocarcinoma | 47
  Moderately differentiated adenocarcinoma | 91
  Poorly differentiated adenocarcinoma | 15
  Mucinous adenocarcinoma | 3
  Other | 8
Information on Primary Lesion: Single, Multiple or Unknown [Count of Participants; unit: Participants]
  Single | 120
  Multiple | 4
  Unknown | 40
Information on Primary Lesion: Primary Lesion Site [Count of Participants; unit: Participants] — Population: Primary tumor location data was collected/analyzed for 124 participants with multiple choices allowed, and total 134 data was available.
  Participants
    Cecum: number analyzed (Participants) | 124
    Cecum | 8
    Ascending colon: number analyzed (Participants) | 124
    Ascending colon | 15
    Transverse colon: number analyzed (Participants) | 124
    Transverse colon | 10
    Descending colon: number analyzed (Participants) | 124
    Descending colon | 4
    Sigmoid colon: number analyzed (Participants) | 124
    Sigmoid colon | 43
    Rectosigmoid: number analyzed (Participants) | 124
    Rectosigmoid | 12
    Rectum: number analyzed (Participants) | 124
    Rectum | 42
History of Surgery [Count of Participants; unit: Participants]
  Had No History of Surgery | 51
  Had History of Surgery | 113
History of Radiotherapy [Count of Participants; unit: Participants]
  Had No History of Radiotherapy | 163
  Had History of Radiotherapy | 1
History of Preoperative and/or Postoperative Adjuvant (Adj) Chemotherapy (CT) [Count of Participants; unit: Participants]
  Had No History of Pre/Postoperative Adj CT | 151
  Had History of Pre/Postoperative Adj CT | 13
Number of Metastatic Organs at Enrollment [Count of Participants; unit: Participants]
  0 | 3
  1 | 72
  ≥2 | 89
Type of Metastatic Organs at Enrollment [Count of Participants; unit: Participants]
  Liver | 119
  Lung | 57
  Peritoneum | 28
  Lymph node | 60
  Bone | 9
  Adrenal gland | 2
  Other | 13
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Cycle 1] [Count of Participants; unit: Participants] — ECOG assessed participant's performance status on 5 point scale: 0=Fully active/able to carry on all pre-disease activities without restriction; 1=restricted in physically strenuous activity but ambulatory/able to carry out light or sedentary work; 2=ambulatory (>50 percent of waking hours), capable of all self-care but unable to carry out any work activities; 3=capable of only limited self-care, confined to bed/chair >50 percent of waking hours; 4=completely disabled, cannot carry on any self-care, totally confined to bed/chair.
  Participants
    0 | 122
    1 | 42
Neuroblastoma Rat Sarcoma (NRAS) + Kirsten Rat Sarcoma (KRAS) Testing [Count of Participants; unit: Participants]
  Mutant-type | 10
  Wild Type (WT) | 152
  Unknown | 2
Worst Grade of Laboratory Tests/Clinical Findings During Protocol Treatment 1 [Count of Participants; unit: Participants] — Grade of Laboratory Tests/Clinical Findings was evaluated based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 4.03 as follows: Grade 1 (mild); Grade 2 (moderate); Grade 3 (severe or medically significant but not immediately life threatening); Grade 4 (life-threatening consequences); Grade 5 (death related to Adverse Events (AE)).
  Participants
    None | 103
    Grade 2 | 21
    Grade ≥3 | 40
Worst Grade of Peripheral Neuropathy During Protocol Treatment 1 [Count of Participants; unit: Participants] — Grade of Peripheral Neuropathy was evaluated based on NCI CTCAE version 4.03 as follows: Grade 1 (mild); Grade 2 (moderate); Grade 3 (severe or medically significant but not immediately life threatening); Grade 4 (life-threatening consequences); Grade 5 (death related to AE).
  Participants
    None | 100
    Grade 1 | 51
    Grade 2 | 12
    Grade ≥3 | 1
Number of Participants without Curative Resection During Protocol Treatment 1 [Count of Participants; unit: Participants] | 164
Treatment Status for Protocol Treatment 1: Reduced or Not Reduced [Count of Participants; unit: Participants] — Treatment status was defined based on a presence or absence of any dose reduction.
  Participants
    Reduced | 59
    Not Reduced | 105
Treatment Status for Protocol Treatment 1: Postponed or Not Postponed [Count of Participants; unit: Participants] — Treatment status was defined based on a presence or absence of any dose delays.
  Participants
    Postponed | 121
    Not Postponed | 43

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival Rate (PFS Rate) at 9 Months After Randomization
Description: PFS rate was defined as the gross percentage of participants who survived with no evidence of progression from the day of randomization (Day 0) until 9 months after Day 0. The presence/absence of progressive disease (PD) was determined based on imaging, consideration of clinical PD, or survival research results. PD based on response evaluation criteria in solid tumors (RECIST) is at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Up to 9 months after randomization
Population: Full Analysis Set (FAS) was defined as all randomized participants.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 56 | 57
percentage of participants | 46.4 [38.1 to 54.9] | 47.4 [39.1 to 55.8]
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; Difference of PFS rate between groups = 0.9, 95% CI 2-sided [-17.2 to 19.0]; Agresti-Caffo method was used for estimation of 95% CI

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: The PFS is the period from the date of randomization (Day 0) until the date of judgment of progression from the date of randomization, or until death by all causes, whichever comes first. The presence/absence of progressive disease (PD) was determined based on imaging, consideration of clinical PD, or survival research results. PD based on response evaluation criteria in solid tumors (RECIST) is at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Up to approximately 31 months
Population: FAS was defined as all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group A | Group B
Number analyzed (Participants) | 56 | 57
months | 9.1 [8.6 to 11.1] | 9.3 [6.0 to 13.0]
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = 0.7349, Regression, Multivariable Cox; The Cox regression model was adjusted by stratification factors except for study sites; Adjusted Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.60 to 1.43]

3. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the day of randomization (Day 0) until death by all causes.
Time Frame: Up to approximately 31 months
Population: FAS was defined as all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group A | Group B
Number analyzed (Participants) | 56 | 57
months | NA [NA to NA] — Median and upper and lower limits of overall survival is not estimable at final analysis due to low number of participants with events. | NA [NA to NA] — Median and upper and lower limits of overall survival is not estimable at final analysis due to low number of participants with events.
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = 0.3485, Regression, Multivariable Cox; The Cox regression model was adjusted by stratification factors except for study sites; Adjusted Hazard Ratio (HR) = 1.41, 95% CI 2-sided [0.69 to 2.88]

4. Secondary Outcome: Response Rate (RR)
Description: RR was defined as the percentage of participants who had shown complete response (CR) or partial response (PR) as the best overall response in accordance with the RECIST 1.1 criteria after randomization. The best overall response was CR, followed by PR, stable disease (SD), progressive disease (PD), and not evaluable (NE). CR: disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to <10 mm. PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters as the best overall response after randomization., SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study).
Time Frame: Up to approximately 31 months
Population: FAS was defined as all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 56 | 57
percentage of participants | 80.4 [68.0 to 88.8] | 87.7 [76.4 to 94.2]

5. Secondary Outcome: Time to Treatment Failure (TTF)
Description: TTF was defined as the time from the day of randomization (Day 0) until the day of protocol treatment discontinuation determination, the day of PD decision during protocol treatment, or death from any cause, whichever came the earliest.
Time Frame: Up to approximately 31 months
Population: FAS was defined as all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group A | Group B
Number analyzed (Participants) | 56 | 57
months | 8.1 [5.9 to 9.5] | 6.1 [4.5 to 9.3]
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = 0.5901, Regression, Multivariable Cox; The Cox regression model was adjusted by stratification factors except for study sites; Multivariable Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.60 to 1.33]

6. Secondary Outcome: Percentage of Participants With Adverse Events
Description: Safety population was defined as all participants who received at least one dose of protocol treatment after randomization.
Time Frame: Up to 28 days after discontinuation of study drug or start of subsequent therapy (data cut off: 31 August 2017; Overall study completion date)
Population: Safety population was defined as all participants who received at least one dose of protocol treatment after randomization.
Measure: Number; unit: percentage of participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 56 | 54
percentage of participants | 100 | 100

7. Secondary Outcome: Percentage of Participants With Adverse Events by Severity Graded Using the Common Terminology Criteria for Adverse Events (CTCAE) Grade
Description: An AE is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medical treatment or procedure that may or may not be considered related to the medical treatment or procedure. Grade refers to the severity of the AE. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 56 | 54
percentage of participants
  Grade 1 | 0 | 0
  Grade 2 | 19.6 | 27.8
  Grade 3, 4 and 5 | 80.4 | 72.2

8. Secondary Outcome: Percentage of Participants With Grade 2 or Higher Peripheral Neuropathy
Description: Peripheral neuropathy was defined as events classified with a preferred term (PT) of "peripheral neuropathy" according to Standardized MedDRA Queries.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 56 | 54
percentage of participants | 30.4 [19.8 to 43.4] | 3.7 [0.3 to 13.3]

9. Secondary Outcome: Percentage of Participants With Grade 3 or Higher Skin Toxicity
Description: Skin toxicity was defined as events classified with an system organ class of "Skin and subcutaneous tissue disorders" or a preferred term of "paronychia".
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 56 | 54
percentage of participants
  Skin and subcutaneous tissue disorders | 17.9 | 18.5
  Paronychia | 7.1 | 9.3

ADVERSE EVENTS:
Time Frame: Up to approximately 34 months
Description: At each visit the investigators had to record any occurrence of adverse events. Adverse events were any unfavorable or unintended sign (including clinically problematic abnormalities of laboratory test data), symptoms, or diseases that developed after the administration of a drug, irrespective of whether there was a causal relationship with the relevant treatment. Safety population included participants who received at least one dose of protocol treatment after randomization.
Arm/Group | Group A | Group B
All-Cause Mortality (participants affected / at risk) | 2/56 | 0/54
Serious Adverse Events (participants affected / at risk) | 20/56 | 18/54
Other Adverse Events (participants affected / at risk) | 47/56 | 45/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=56) | Group B (N=54)
Mechanical ileus (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Device related infection (Infections and infestations) | 2 | 0
Pelvic abscess (Infections and infestations) | 0 | 1
Biliary tract infection (Infections and infestations) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Chest discomfort (General disorders) | 1 | 0
Death (General disorders) | 1 | 0 — One treatment emergent death occurred during the treatment and is related to treatment.
Pyrexia (General disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 — One treatment emergent death occurred during the treatment and is related to treatment.
Cholangitis (Hepatobiliary disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0
Nutritional condition abnormal (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 1
Enteritis infectious (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Amylase increased (Investigations) | 0 | 1
Heat illness (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Embolism (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=56) | Group B (N=54)
Neutrophil count decreased (Investigations) | 18 (44) | 15 (19)
White blood cell count decreased (Investigations) | 7 (12) | 9 (18)
Platelet count decreased (Investigations) | 5 (17) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 8 (8) | 6 (6)
Dysgeusia (Nervous system disorders) | 7 (7) | 4 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3) | 3 (3)
Paronychia (Infections and infestations) | 14 (14) | 16 (16)
Hypomagnesaemia (Metabolism and nutrition disorders) | 10 (10) | 11 (12)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5) | 4 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (4)
Stomatitis (Gastrointestinal disorders) | 5 (5) | 5 (6)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (4)
Vomiting (Gastrointestinal disorders) | 4 (7) | 1 (1)
Malaise (General disorders) | 4 (5) | 4 (4)
Pyrexia (General disorders) | 4 (4) | 3 (3)
Fatigue (General disorders) | 3 (3) | 0 (0)
Hypersensitivity (Immune system disorders) | 6 (8) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-12-20): https://cdn.clinicaltrials.gov/large-docs/46/NCT02337946/SAP_000.pdf
  • Study Protocol (2016-10-20): https://cdn.clinicaltrials.gov/large-docs/46/NCT02337946/Prot_001.pdf